CLINICAL TRIAL: NCT03852238
Title: Risk Factors of Hepatocellular Carcinomas Developed on Non-fibrotic Liver (NoFlic Study)
Brief Title: Risk Factors of Hepatocellular Carcinomas Developed on Non-fibrotic Liver: Case-control Study (NoFlic Study)
Acronym: NoFlic
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2010/03
Record Dates: First submitted 2019-01-31; First posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; Non-cirrhotic liver; Risk factors
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: patients with hepatocellular carcinoma on non-cirrhotic: Blood test and self-administrated questionnaires (medical history of the participant and his / her family, tobacco consumption, alcoholic and non-alcoholic beverages consumption, eating habits, type of employment and exposure, stays abroad longer than 1 month
- Control: patients without hepatocellular carcinoma: Blood test and self-administrated questionnaires (medical history of the participant and his / her family, tobacco consumption, alcoholic and non-alcoholic beverages consumption, eating habits, type of employment and exposure, stays abroad longer than 1 month
  Interventions: Other: Blood test and self-administrated questionnaires

INTERVENTIONS:
Other: Blood test and self-administrated questionnaires
  Groups: Control: patients without hepatocellular carcinoma

SUMMARY:
The main objective of this study is to identify direct carcinogenic factors in the absence of cirrhosis, and the carcinogenesis pathways involved on nonfibrotic liver (NfCHC).

DETAILED DESCRIPTION:
Most hepatocellular carcinoma (HCC) complicates cirrhosis, which is often caused by infection with hepatitis B or C viruses, alcohol, obesity, exposure to aflatoxin B1 (AFB1) or hemochromatosis. Nevertheless, 10 to 40% of HCCs can develop on non-cirrhotic terrain and about 5% on nonfibrotic liver (NfHCC). In 20 to 40% of these NfHCCs, no classical HCC risk factor is identified. Some cases could be the result of a transformation of an adenoma. Others may be associated with yet non-formally identified toxins and / or a specific genetic predisposition. While there is a lot of data on alterations of signaling pathways (ß-catenin, AKT / mTOR, Ras / pERK, etc.) in "classical" HCCs, altered pathways remain unknown in most NfHCCs, even in some cases, activation of β-catenin, inactivating mutations of HNF1 or activators of gp130 have been shown. A specific study of NfHCCs, rather rare cancers, represents an opportunity to look for directly carcinogenic factors in the absence of cirrhosis, and to dissect the involved carcinogenesis pathways.

ELIGIBILITY:
Inclusion Criteria:

* CASES: patients aged 18 years and older with a diagnosis of NfHCC with anatomopathological examination and showing a HCC according to standard histopathological criteria and an absence of significant fibrosis in non-tumoral tissues with the METAVIR system score or equivalent (F0 or F1) or the Kleiner et al stage of ASH and NASH (≤stade 2); signed informed consent; affiliated or beneficiary of a social security system
* CONTROLS: patients aged 18 years and older without NfHCC at baseline; patients for whom an endoscopy is programmed as part of an assessment of intestinal functional disorders, dyspeptic disorders or screening colonoscopy or hospitalized patients in orthopedic surgery / traumatology or rheumatology departments; signed informed consent; affiliated or beneficiary of a social security system

Exclusion Criteria:

* CASES: HCC diagnosed without pathological examination; hepatic transplantation before the diagnosis of HCC; patients unable to answer questions; patients who do not speak French or live abroad.
* CONTROLS: History of liver cancer; other cancers under treatment except cutaneous cancers; Colonoscopy indicated in case of familial form of colon cancer; patient with cirrhosis; patients unable to answer questions; patients who do not speak French or live abroad; Relationship or same home with the case

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CASES: patients with a diagnosis of NfHCC with anatomopathological examination and showing a HCC according to standard histopathological criteria and an absence of significant fibrosis in non-tumoral tissues with the METAVIR system score or equivalent (F0 or F1) or the Kleiner et al stage of ASH and NASH (≤stade 2)
  - CONTROLS: patients without NfHCC at baseline
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2010-08-18 (Actual); Primary Completion 2013-11-14 (Actual); Study Completion 2013-11-14 (Actual)

PRIMARY OUTCOMES:
exposure to Viral hepatitis B | Baseline
  binary yes / undiagnosed by positive serology for anti-HBc antibodies isolated or associated with positive serology for anti-HBs antibodies

SECONDARY OUTCOMES:
exposure to viral hepatitis C | baseline
  binary yes / undiagnosed by positive serology for positive anti-HCV antibodies

OTHER OUTCOMES:
exposure to Alcohol | baseline
  binary variable, separating large consumers from others
exposure to Exogenous female hormones | baseline
  oral contraceptive coded as a binary variable
history of liver pathology | baseline
  binary variable: yes/no
Family history of liver cancer | baseline
  binary variable: yes/no
Diabetes | baseline
  categorical variable (depending on the type of diabetes: 1 or 2).
Dyslipidemias | baseline
  qualitative variables: hypercholesterolemia / hyper triglyceridemia
Medical treatments for dyslipidemia | baseline
  depending on the type of medication: statins, fibrates, other
Metabolic syndrome | baseline
  binary variable: present / absent
Age of first menstruation | baseline
  quantitative variable in years
Parity | baseline
  number of children
breastfeeding | baseline
  binary variable : yes / no
Menstrual status | baseline
  menopausal status will be treated as a binary variable
Duration of exposure to different variables | baseline
  quantitative variable in months
fruits | baseline
  frequency of intake assessed by a frequency food questionnaire
vegetables | baseline
  frequency of intake assessed by a frequency food questionnaire
meat | baseline
  frequency of intake assessed by a frequency food questionnaire
fish | baseline
  frequency of intake assessed by a frequency food questionnaire
dairy products | baseline
  frequency of intake assessed by a frequency food questionnaire
fats | baseline
  frequency of intake assessed by a frequency food questionnaire

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - CHU Amiens, Amiens
  - AP-HP Jean Verdier, Bondy
  - CHU Bordeaux, Bordeaux
  - CHU Caen, Caen
  - AP-HP Hopital Antoine Béclère, Clamart
  - AP-HP Hopital Beaujon, Clichy
  - CHI Créteil, Créteil
  - CHU Grenoble, Grenoble
  - Hopital Edouard Herriot, Lyon
  - Hospices Civiles de Lyon, Lyon
  - AP-HP Cochin, Paris
  - AP-HP Hopital Henri Mondor, Paris
  - AP-HP Hopital Saint Antoine, Paris
  - CHU Villejuif, Villejuif

IPD SHARING:
Plan to Share IPD: No